CLINICAL TRIAL: NCT02262221
Title: Health and Economic Outcomes of Two Different Follow up Strategies in Effectively Cured Advanced Head and Neck Cancer
Acronym: HETeCo
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Low participant accrual
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Bocconi University (Other); University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: INT 48/14
Record Dates: First submitted 2014-10-06; First posted 2014-10-13 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A (Non intensive Follow up) (No Intervention): Follow up consisting of outpatient visits according to the schedule foreseen for single head and neck subsite. At each follow up visit patients will report all new symptoms and they will receive physical and fiberoptic endoscopic head and neck examination. Laboratory tests will be performed once a year. Quality of life questionnaires will be administered to patients every other visit for the first 2 years and then at each visit. A socio-economic questionnaire will be also administered at each visit. Locoregional imaging will be performed within 6 months after radiotherapy end and recommended only at the occurrence of new signs or symptoms. Patients will be contacted by a phone call between visits in order to monitor patient's reported symptoms potentially related to disease recurrence.
- ARM B (Intensive Follow up) (Other): Intervention foreseen is scheduled radiologic evaluations (CT or MRI scan) and PET scan if patients ≥ 50 years old and with a smoking history ≥ 20 pack year. Follow up outpatient visits will be performed similarly to ARM A, including physical and fiberoptic endoscopic head and neck evaluation and laboratory tests and questionnaires. Locoregional imaging will be requested for all the patients 2 times/year in the first 2 years and 1 time/year in the third and fourth year; PET scan will be requested yearly in the first 3 years. In the first year after RT end, MRI or CT scan will be performed at screening and at sixth month after enrollment, while PET scan will be performed six months after enrollment only in patients ≥50 years and with a smoking history of ≥20 pack/years.
  Interventions: Other: Scheduled radiologic evaluations

INTERVENTIONS:
Other: Scheduled radiologic evaluations — Scheduled radiologic evaluations (CT or MRI scan) and PET scan in the case that patiets are ≥ 50 years old and with a smokink history ≥ 20 pack year
  Arms: ARM B (Intensive Follow up)

SUMMARY:
Randomized, multicenter trial to evaluate the cost-effectiveness of 2 different follows up programs in head and neck cancer survivors. Patients in complete remission at month 6 (+/- 1 month) after curative treatment will be randomized in two arms according to 2 different follow up approaches: Non Intensive Follow up approach (Arm A) with no radiologic evaltuations scheduled, but required only at the occurence of any signs or symptoms and Intensive Follow up approach (Arm B) with scheduled radiologic evaluations.

DETAILED DESCRIPTION:
The choice about timing of follow visits for each patient will be performed before randomization and will be tailored to the single patient in accordance to NCCN and AIOCC guidelines following this scheduling:

* Oral Cavity cancer: every 2 months for the 1st year, every 3 months in the 2nd year, every 4 months in the 3rd year and every 6 months in the 4th and 5th year
* Oropharyngeal and laryngeal cancer: every 3 months for the 1st and the 2nd year, every 4 months in the 3rd year and every 6 months in the 4th and 5th year
* Hypopharyngeal cancer: every 3 months for the 1st and the 2nd year, every 6 months from the 3rd to the 5th year

Patients deemed to be in complete remission at month 6 (+/- 1 month) after curative treatment will be randomized in two follow up arms:

ARM A (Non intensive): follow up according to NCCN guidelines, consisting of outpatient visits according to the schedule foreseen for single head and neck subsite. At each follow up visit the patients will report all new symptoms and they will receive both physical and fiberoptic endoscopic head and neck examination.

Laboratory tests (complete blood count, renal, hepatic and thyroid function) will be performed once a year. Quality of life questionnaire (EuroQol 5D5L, EORTC QLQ C-30 and HN35) will be administered to patients every other visit for the first 2 years and then at each visit. During each visit, a socio-economic questionnaire will be also administered. Locoregional imaging will be performed within 6 months after treatment end and then will be recommended only on the occurrence of new signs or symptoms. Only patients in this arm will be contacted by a phone call between visits in order to monitor patient's reported symptoms which could be potentially related to disease recurrence.

ARM B (Intensive): follow up outpatient visits will be performed similarly to ARM A, including physical and fiberoptic endoscopic head and neck evaluation and laboratory tests and questionnaires. Locoregional imaging will be requested for all the patients 2 times/year in the first 2 years and 1 time/year in the third and fourth year; PET scan will be requested yearly in the first 3 years.

In the first year after RT end, MRI or CT scan will be performed at screening and at sixth month after enrollment, while PET scan will be performed six months after enrollment. Radiological imaging with PET will be customized according to smoking history being performed in subjects >50 years and with a smoking history of > 20 pack/years.

Randomization will be stratified according to site of primary disease, smoking history (> 10pack years) and likelihood of feasibility or non feasibility of salvage surgery if a recurrence at T/N level would emerge (salvage surgery feasibility).

ELIGIBILITY:
Inclusion Criteria:

* Clinical or pathological stage III-IV squamous cell head and neck cancer of oral cavity, oropharynx, larynx or hypopharynx after curative treatment
* Oropharyngeal cancer will be enrolled only if HPV negative or HPV positive with a smoking history (i.e. greater than 10 packs/year)
* Having already received Radiation Therapy (RT) as curative treatment or in postoperative setting
* Patients without evidence of disease within six months after treatment end (first assessment of disease must be performed with radiological imaging for all patients)
* Patient randomization must be performed at the sixth month after RT end (+/- 1 month)
* Patients having or not received systemic treatment for a curable disease are allowed
* Patients not considered suitable for salvage surgery (based on primary tumor characteristics and previous treatments) after hypothetical recurrence are allowed; the choice about feasibility or non feasibility of salvage surgery in case of hypothetical recurrence at T or N level will be made by the multidisciplinary team before randomization (salvage surgery score)
* 18 years or older
* Informed consent signed

Exclusion Criteria:

* Patient with primary tumor site: nasopharynx, paranasal sinus, salivary gland or with cancer of unknown primary in head and neck district
* Patients unable to comply with the protocol, in the opinion of the investigator
* Any other malignancy (except for appropriately treated superficial basal cell skin cancer and surgically cured cervical cancer in situ) unless free of disease for at least five years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2014-06; Primary Completion 2020-07 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the most cost-effective follow up strategy | 3 years
  To evaluate the most cost-effective follow up strategy by comparing health consequences and costs of the two alternative follow-up strategies.

SECONDARY OUTCOMES:
Evaluation of the percentage of potentially salvageable recurrences or second primaries | 3 years
  To evaluate the percentage of potentially salvageable recurrences or second primaries in both groups of follow up approach.
Assessment of the cause-specific survival | 3 years
  To assess the cause-specific survival (CSS).
Assessment of the OS of patients recurring | 3 years
  To assess the overall survival (OS) of patients recurring in both groups of follow up approach.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Licitra, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (15):
- Italy (13):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milano, Milan, MI
  - Policlino S. Orsola-Maplighi, Bologna
  - Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Istituto Nazionale per la ricerca sul cancro, Genova
  - Istituto Europeo di Oncologia, Milan
  - Policlinico di Modena, Modena
  - Istituto Nazionale Tumori IRCCS - Fondazione Pascale, Napoli
  - Ospedale di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Santa Maria degli Angeli, Pordenone
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Ospedale di Trento, Trento
- Switzerland (2):
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - CHUV - Centre hospitalier universitaire vaudois, Lausanne

IPD SHARING:
Plan to Share IPD: Yes
Study results will be shared trough pubblications, abstracts and posters

REFERENCES:
- [Derived] Meregaglia M, Cairns J, Licitra L, Bossi P. The use of intensive radiological assessments in routine surveillance after treatment for head and neck cancer: An economic evaluation. Eur J Cancer. 2018 Apr;93:89-98. doi: 10.1016/j.ejca.2018.01.082. Epub 2018 Mar 20. PMID 29477796